CLINICAL TRIAL: NCT02935959
Title: Premedication With Different Nebulized Ketamine,Dexmedetomidine Versus Midazolam in Oncologic Preschool Children
Brief Title: Premedication With Nebulized Ketamine,Dexmedetomidine Versus Midazolam in Oncologic Preschool Children
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shereen Mamdouh, lecturer of anesthesia,ICU and pain management, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 349
Record Dates: First submitted 2016-10-12; First posted 2016-10-18 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Oncological Children

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- nebulized ketamine (Active Comparator): patients will be premedicated with nebulized ketamine solution (2 mg/kg)
  Interventions: Drug: nebulized ketamine
- nebulized dexmedetomidine (Active Comparator): patients will be premedicated with nebulized dexmedetomidine solution (2 μg/kg)
  Interventions: Drug: nebulized Dexmedetomidine
- nebulized midazolam (Active Comparator): patients will be premedicated with midazolam (0.2 mg/kg) nebulized solution
  Interventions: Drug: nebulized midazolam

INTERVENTIONS:
Drug: nebulized ketamine — Drugs will be prepared in 3 mL of saline 0.9% before administration by a standard hospital jet nebulizer via a mouthpiece, with a continuous flow of 100% oxygen at 6 L/min for 10 to 15 minutes (30 minutes before GA). Treatment will be stopped when the nebulizer began to sputter.
  Arms: nebulized ketamine
Drug: nebulized Dexmedetomidine
  Arms: nebulized dexmedetomidine
Drug: nebulized midazolam
  Arms: nebulized midazolam

SUMMARY:
Evaluate the efficacy of nebulized dexmedetomidine, nebulized ketamine, and nebulized midazolam a premedication prior to general anesthesia (GA) in oncologic preschool children undergo bone marrow aspirate and biopsy.

DETAILED DESCRIPTION:
The preoperative period can be a traumatic time for young children undergoing surgery. Pediatric anesthesiologists strive to minimize distress for children in the operating room (OR) environment and to provide a smooth induction of anesthesia. Preoperative anxiety stimulates the sympathetic, parasympathetic, and endocrine systems, leading to an increase in heart rate (HR), blood pressure, and cardiac excitability. Various drugs have been advocated as premedication to allay anxiety and facilitate the smooth separation of children from parents. The ideal premedicant in children should be readily acceptable and should have a rapid and reliable onset with minimal side effects. Dexmedetomidine is a tasteless, colorless, and odorless drug that acts as a selective α-2 adrenergic agonist with both sedative and analgesic effects via actions in the central nervous system. Ketamine is an N-methyl-d-aspartate receptor antagonist that produces a state of sedation, anesthesia, immobility, analgesia, amnesia, and dissociation from the environment. Midazolam is a water-soluble benzodiazepine known to have a rapid onset and short duration of action, as well as properties of amnesia and anxiolysis. Administered intranasally, midazolam is an effective option for conscious sedation.

ELIGIBILITY:
Inclusion Criteria:

* physical status I and II, scheduled for bone marrow aspirate and biopsy

Exclusion Criteria:

* known allergy to the studied drugs,
* organ dysfunction,
* cardiac dysrrhythmia and/or congenital heart disease,
* psychotropic medication use and mental retardation

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2016-10; Primary Completion 2017-09 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
the degree of sedation when the child was first seen in the OR | 30 minutes after sedation
  measure the degree of sedation using using a 5 point sedation scale. Sedation level: Agitated =1, alert= 2, calm= 3, drowsy = 4, asleep=5.

SECONDARY OUTCOMES:
parental separation | 30 min after sedation
  The parental separation anxiety scale (PSAS)
Emergecy agitation | 30 min after induction
  Emergence agitation will be assessed according to a 3-point scale: 1 = calm; 2 = restless but calms to verbal instructions; and 3 = combative and disoriented.

CONTACTS AND LOCATIONS:
Overall Officials: fatma a elsherif, lecturer, Study Chair — South Egypt Cancer Institute
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Derived] Abdel-Ghaffar HS, Kamal SM, El Sherif FA, Mohamed SA. Comparison of nebulised dexmedetomidine, ketamine, or midazolam for premedication in preschool children undergoing bone marrow biopsy. Br J Anaesth. 2018 Aug;121(2):445-452. doi: 10.1016/j.bja.2018.03.039. Epub 2018 Jun 22. PMID 30032884